CLINICAL TRIAL: NCT05320926
Title: Clopidogrel Versus Aspirin MOnotherapy After 1- to 3-month of Dual-antiplatelet thErapy Following Zotarolimus-eluting Onyx Stents Implantation; C-MODE Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2022-0050
Record Dates: First submitted 2022-04-03; First posted 2022-04-11 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-term DAPT followed by clopidogrel monotherapy (Experimental): atients who received zotarolimus-eluting Onyx stents implantation for treating ischemic heart disease at de novo coronary lesion will maintain 1-3 months DAPT. Patients will be randomized to stop aspirin and maintain clopidogrel after DAPT.
  Interventions: Drug: Clopidogrel monotherapy; Device: zotarolimus-eluting stent (Resolute Onyx ®)
- Short-term DAPT followed by aspirin monotherapy (Active Comparator): Arm Description: Patients who received zotarolimus-eluting Onyx stents implantation for treating ischemic heart disease at de novo coronary lesion will maintain 1-3 months DAPT. Patients will be randomized to stop clopidogrel and maintain aspirin after DAPT.
  Interventions: Drug: Aspirin monotherapy; Device: zotarolimus-eluting stent (Resolute Onyx ®)

INTERVENTIONS:
Drug: Clopidogrel monotherapy — Patients will be randomized to stop aspirin and maintain clopidogrel after short-term DAPT.
  Arms: Short-term DAPT followed by clopidogrel monotherapy
Drug: Aspirin monotherapy — Patients will be randomized to stop clopidogrel and maintain aspirin after short-term DAPT.
  Arms: Short-term DAPT followed by aspirin monotherapy
Device: zotarolimus-eluting stent (Resolute Onyx ®) — zotarolimus-eluting stent (Resolute Onyx ®)

SUMMARY:
Previous randomized clinical trials have deomonstrated the efficacy and safety of short-term dual antiplatelet therapy (DAPT) after percutaneous coronary intervention (PCI), however, the single antiplatelet agent to be maintained after short-term DAPT was different. Therefore, which antiplatelet agent to be maintained after short-term DAPT needs further invstigations.

DETAILED DESCRIPTION:
The investigators hypothesized that short-term (1-3 months) DAPT followed by clopidogrel monotherapy will be superior to short-term DAPT followed by aspirin monotherapy after PCI in patients with ischemic heart disease. We will evaluate whether clopidogrel monotherapy will reduce the rate of net adverse clinical events (NACE) at 12 months compared to aspirin monotherapy after very-short term DAPT. Eligible patients will be randomized to short-term DAPT followed by clopidogrel monotherapy or short-term DAPT followed by aspirin monotherapy at hospitalization for index PCI. Randomization will be stratified according to 1) bleeding risk (high bleeding risk [HBR] or non-HBR), 2) clinical presentation (acute coronary syndrome or chronic coronary artery disease), and 3) lesion complexity (non-complex or complex lesion). Regarding the duration of very-short term DAPT, the maintenance duration of DAPT (1-month or 3-month) will be determined as follows:

* If the patients are at HBR (HBR is defined according to ARC-HBR criteria: meeting at least 1 major or 2 minor criteria), 1-month DAPT will be given regardless of clinical presentation or lesion complexity.
* In the patients are at non-HBR, 3-month DAPT will be given in those treated for unstable angina and/or complex lesions (complex lesion is defined as meeting at least one of the following: number of stents implanted ≥3, number of lesions treated ≥3, 3-vessel treated, bifurcation PCI with 2 stents, total stent length ≥60mm, or chronic total occlusion).

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥19 years
2. Patients who received new generation zotarolimus-eluting Onyx stents implantation for treating ischemic heart disease
3. Provision of informed consent

Exclusion Criteria:

1. Age ≥ 85 years
2. Acute myocardial infarction

2. Left main bifurcation requiring 2-stent technique 3. Pregnant women or women with potential childbearing 4. Life expectancy < 1 year 5. Inability to follow the patient over the period of 1 year after enrollment, as assessed by the investigator 6. Inability to understand or read the informed consent

Ages: 19 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3744 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2028-07-10 (Estimated); Study Completion 2028-07-10 (Estimated)

PRIMARY OUTCOMES:
Net adverse clinical events (NACE) | 1 year after the procedure
  Composite of all-cause death, myocardial infarction, stroke, or major bleeding (BARC 2, 3 or 5)

SECONDARY OUTCOMES:
Each component of NACE | 1 year after the procedure
Major adverse cardiac and cerebrovascular events (MACCE: composite of all-cause death, myocardial infarction, or stroke) | 1 year after the procedure
Cardiac death | 1 year after the procedure
Stent thrombosis (definite or probable) | 1 year after the procedure
Target-vessel revascularization | 1 year after the procedure
Target-lesion revascularization | 1 year after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Byeong-Keuk Kim, Principal Investigator — Severance Cardiovascular Hospital, Yonsei University Health System
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No